CLINICAL TRIAL: NCT06273800
Title: Chemosensitivity During Phases of the Menstrual Cycle in Breast Cancer Patients
Acronym: Chemosense
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M23CMC
Record Dates: First submitted 2024-02-15; First posted 2024-02-23 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Triple negative tumor; Stage I - III disease; Starting neo adjuvant treatment; Regular physiological menstrual cycle (premenopausal)
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: collection of serum sample blood at first day of neo adjuvant treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sample (Other): Collection of serum blood sample at day of start neo adjuvant treatment
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — Collection of serum sample at the day of start of neo adjuvant treatment

SUMMARY:
This study is a prospective, multicenter study in which a serum sample will be collected at the day of starting neo adjuvant treatment in breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

* Women with a new diagnosis of triple negative breast cancer who have not yet started systemic treatment.
* Patients with stage I-III disease, patient with locoregional recurrence who have not been treated with chemotherapy before. ,
* Aged < 60 years
* Women having a (regular) physiological menstrual cycle
* Patients who are assigned to receive neoadjuvant chemotherapy with or without immunotherapy, targeted therapy and endocrine therapy
* Patients must be systemic treatment naïve for current malignancy (e.g. no chemotherapy, hormonal therapy or targeted therapy)
* Signed written informed consent

Exclusion Criteria:

* current use of hormonal contraception or in the six weeks prior to start of neoadjuvant systemic treatment for breast cancer, such as:
* Oral contraception (OAC)
* Hormonal intra-uterine device (IUD, Mirena)
* No ovarian function suppression to preserve fertility
* Other forms of hormonal contraception, including but not limited to: nuva-ring, Implanon, prikpil
* Currently pregnant and / or breast feeding. In case of use of hormonal contraception or breast feeding in de last year: patients should have had at least 2 menstrual cycles since stopping hormonal contraception.

  - active other malignancy
* IVF-trajectory for egg cell preservation prior to start of neoadjuvant systemic treatment

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2035-07-15 (Estimated); Study Completion 2036-07-15 (Estimated)

PRIMARY OUTCOMES:
pCR rate | At 6 months
  Number of patients achieving a pathological complete response

SECONDARY OUTCOMES:
Radiological reduction on tumor size | At 6 months
  Number of patients achieving a radiological response (CR, PR, SD) based on MRI after neo adjuvant treatment
Pathological reduction on tumor size | At 6 months
  Number of patients achieving a pathological response (CR, PR, SD) based on pathology report after neo adjuvant
Residual cancer burden (RCB) | At 6 months
  quantificaton of the residual disease after neoadjuvant therapy
Distant recurrence free interval (DRFI) | Up to 120 months
  Number of patients with distant recurrence
Recurrence-free interval (RFI) | Up to 120 months
  Number of patients with disease recurrence
Overall survival (OS) | Up to 120 months
  Number of patients alive or deceased

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Linn, MD, Principal Investigator — Antoni van Leeuwenhoek
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
will follow